CLINICAL TRIAL: NCT05913024
Title: A Single-center, Randomized, Blinded, Different Doses, Positive Control, Phase II to Evaluate the Inactivated EV71 Vaccine Immunogenicity and Safety in Healthy Volunteers Aged 6 to 71 Months
Brief Title: Immunogenicity and Safety of Enterovirus Type 71 Vaccine,Inactivated(Vero Cells) in Volunteers Aged From 6 to 71 Months
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing Zhifei Lvzhu Biopharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 202101025
Record Dates: First submitted 2023-06-12; First posted 2023-06-22 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-07

CONDITIONS: Healthy Volunteers
Keywords: Enterovirus Type 71 Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Enterovirus Type 71 Vaccine,Inactivated(Vero Cells),high dose (Experimental): Participants received two doses of the vaccine, 28 days apart
  Interventions: Biological: Enterovirus Type 71 Vaccine
- Enterovirus Type 71 Vaccine,Inactivated(Vero Cells),low dose (Experimental): Participants received two doses of the vaccine, 28 days apart
  Interventions: Biological: Enterovirus Type 71 Vaccine
- Enterovirus Type 71 Vaccine,Inactivated(Human Diploid Cell) (Active Comparator): Participants received two doses of the vaccine, 28 days apart
  Interventions: Biological: Enterovirus Type 71 Vaccine

INTERVENTIONS:
Biological: Enterovirus Type 71 Vaccine — Participants received two doses of the vaccine, 28 days apart

SUMMARY:
The goal of this clinical trial is to evaluate the immunogenicity and safety of Enterovirus Type 71 Vaccine,Inactivated(Vero Cells) in healthy volunteers aged from 6 to 71 months.

DETAILED DESCRIPTION:
The goal of this clinical trial is to evaluate the immunogenicity and safety of Enterovirus Type 71 Vaccine,Inactivated(Vero Cells) in healthy volunteers aged from 6 to 71 months.

Qualified subjects were screened and randomly divided into low-dose group, high-dose group, and control group according to the ratio of 2:2:1. The experimental group was vaccinated with the experimental vaccine (low-dose or high-dose enterovirus 71 inactivated vaccine from Beijing Zhifei Lvzhu Biopharmaceutical Co., Ltd.), and the control group was vaccinated with the control vaccine (enterovirus 71 inactivated vaccine produced by the Institute of Medical Biology of the Chinese Academy of Medical Sciences). All participants received two doses of the vaccine 28 days apart.

ELIGIBILITY:
Inclusion Criteria:

* Age 6-71 months, valid identification;
* Infants aged 6-11 months should be full-term (37-42 weeks gestation) and have a birth weight (2500g≤ weight ≤4000g);
* The subject's guardian voluntarily consented to the child's participation in the study and signed an informed consent form;
* The subject's guardian had the ability to learn about the study procedure and was able to participate in all planned follow-ups;
* Pre-enrollment axillary body temperature < 37.5°C.

Exclusion Criteria:

* Have received any previous HFMD vaccine;
* Previous history of hand, foot and mouth disease；
* History of allergies to any component of the study vaccine or substances used in the preparation process，or a history of severe adverse effects of vaccine/drug；
* Have a serious congenital malformation or chronic medical condition that may interfere with the conduct or completion of the study；
* History of seizures, epilepsy, encephalopathy, and psychosis (including family history)；
* Have contraindications to intramuscular injections such as thrombocytopenia, any coagulopathy, or being treated with anticoagulants；
* Have an infectious disease with clinical or serological evidence；
* Patients with asplenia, splenectomy, or functional asplenia due to any condition；
* Patients with congenital or acquired immunodeficiency; or receive systemic corticosteroids within 3 months prior to enrollment, or be on other immunosuppressants prior to enrollment；
* Have received treatment with blood or blood-related products within 3 months prior to enrollment；
* Have acute illness or are in an acute exacerbation of chronic disease within 3 days prior to the first dose of vaccination, or antipyretic, analgesic, and antiallergic medications have been used；
* Have received any inactivated vaccine within 7 days before the first dose, and any live attenuated vaccine within 14 days prior to vaccination；
* Severely abnormal labor (dystocia at birth, instrumental delivery, excluding caesarean section) or history of asphyxia, neurological damage, IVF or multiple births, pathological jaundice (only for infants 6 to 11 months of age)；
* Those who plan to move before the end of the study visit or who are away from the local area for an extended period of time during the scheduled study visit；
* Ongoing or planned participation in clinical trials of other drugs；
* The investigators considered that the participants had any conditions that might interfere with the assessment of the purpose of the study.

Ages: 6 Months to 71 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 470 (Actual)
Dates: Start 2021-10-19 (Actual); Primary Completion 2022-10-24 (Actual); Study Completion 2022-10-24 (Actual)

PRIMARY OUTCOMES:
Anti-EV71 serum neutralizing antibody positive conversion rate at 28 days after immunization | 28 days after two doses of vaccination
  to evaluate immunogenicity of Enterovirus Type 71 Vaccine
Geometric mean titer (GMT) and growth factor of anti-EV71 serum neutralizing antibody 28 days after immunization | 28 days after two doses of vaccination
  to evaluate immunogenicity of Enterovirus Type 71 Vaccine
Ratio of subjects with anti-EV71 serum neutralizing antibody titer ≥ 1:8 28 days after immunization | 28 days after two doses of vaccination
  to evaluate immunogenicity of Enterovirus Type 71 Vaccine
Adverse events within 0-28 days after each dose of vaccination | 28 days after each dose of vaccination
  to evaluate Safety of Enterovirus Type 71 Vaccine

CONTACTS AND LOCATIONS:
Overall Officials: Du lin, master, Study Chair — Beijing Zhifei Lvzhu Biopharmaceutical Co., Ltd
Locations (1):
- Hunan Provincial Center for Disease Control and Prevention, Changsha, Hunan, China